CLINICAL TRIAL: NCT04287517
Title: Efficacy of Capacitive-Resistive Therapy on the Treatment of Neck/Upper Trapezius Myofascial Pain: A Randomized Double-Blind Placebo-Controlled Study
Brief Title: Efficacy of Capacitive-Resistive Therapy on the Treatment of Myofascial Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Sergen Devran, Principal Investigator, Sports Medicine Residency, Medical Doctor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Capacitive-resistive Therapy
Record Dates: First submitted 2020-02-21; First posted 2020-02-27 (Actual); Results first posted 2020-04-15 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Myofascial Pain Syndrome of Neck
Keywords: Myofascial Neck Pain; Capacitive-resistive Therapy
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Capacitive-Resistive Therapy Group (Active Comparator): This group was treated with capacitive resistive diathermy and exercise
  Interventions: Device: Capacitive-Resistive Therapy
- Sham Group (Sham Comparator): This group was treated with sham capacitive-resistive diathermy and exercise
  Interventions: Device: Capacitive-Resistive Therapy

INTERVENTIONS:
Device: Capacitive-Resistive Therapy — Capacitive-resistive diathermy therapy heats deep tissues by transferring energy through radiofrequency waves.
  Other Names: Exercise

SUMMARY:
Myofascial pain syndrome (MPS) is a painful musculoskeletal condition affecting the individuals' daily life presenting with muscle spasm, referred pain patterns, stiffness, restricted range of motion caused by trigger points. Capacitive-resistive diathermy therapy heats deep tissues by transferring energy through radiofrequency waves. Currently, although this modality is used to treat various acute or chronic musculoskeletal disorders, there is no specific data about myofascial trigger points in the literature. The investigators aimed to evaluate the efficacy of capacitive-resistive diathermy on the myofascial trigger point of neck/upper trapezius muscle area compared with the sham intervention of capacitive-resistive diathermy.

Volunteers with active myofascial trigger points in the upper trapezius and neck were included the study after being examined by sports medicine specialists. Exclusion criteria were fibromyalgia, discal hernia, radiculopathy, myelopathy, having received trigger point injection and physical therapy within the last 1 month, neck or back surgery, rheumatismal diseases, pregnancy. Patients were randomly allocated into two groups. Group 1 will be treated with capacitive resistive diathermy and exercise. Group 2 will be treated with placebo (sham) capacitive-resistive diathermy and exercise for 10 sessions at intervals of 24-48 hours. Visual analog scale (VAS), neck disability index (NDI) score, cervical range of motion (cROM), active trigger point numbers will be evaluated before and after treatment. The study was designed as a prospective, randomized, placebo-controlled double-blind trial. The study was approved by the Istanbul Faculty of Medicine Ethics Committee. All participants were informed of the study and signed written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers
* Active myofascial trigger points in the upper trapezius and neck

Exclusion Criteria:

* Fibromyalgia
* Discal Hernia
* Radiculopathy, Myelopathy
* Having received trigger point injection and physical therapy within the last 1 month
* Neck or Back surgery
* Rheumatismal diseases
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sensu Dincer, Dr., Principal Investigator — Istanbul University Faculty of Medicine Sports Medicine Department
Locations (1):
- Istanbul University Faculty of Medicine Sports Medicine Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Patients do not want to share the data with anyone other than the researchers involved in the study.

REFERENCES:
- [Background] Diego IMA, Fernandez-Carnero J, Val SL, Cano-de-la-Cuerda R, Calvo-Lobo C, Piedrola RM, Oliva LCL, Rueda FM. Analgesic effects of a capacitive-resistive monopolar radiofrequency in patients with myofascial chronic neck pain: a pilot randomized controlled trial. Rev Assoc Med Bras (1992). 2019 Feb;65(2):156-164. doi: 10.1590/1806-9282.65.2.156. PMID 30892438
- [Background] Ong J, Claydon LS. The effect of dry needling for myofascial trigger points in the neck and shoulders: a systematic review and meta-analysis. J Bodyw Mov Ther. 2014 Jul;18(3):390-8. doi: 10.1016/j.jbmt.2013.11.009. Epub 2013 Nov 9. PMID 25042309

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty volunteer patients who had active pain in the neck region for the last 1 month, who applied to our clinic (Istanbul University Faculty of Medicine Sports Medicine Department), between 12 December 2019 - 01 March 2020, and who had an active myofascial trigger point were evaluated and included in the study.
Pre-assignment Details: Although 2 patients met the diagnostic criteria, they were not included in the study due to cervical hernia and cervical stenosis.
Period: Overall Study
Arm/Group | Capacitive-Resistive Therapy Group | Sham Group
Started | 19 | 19
Completed | 18 | 18
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Capacitive-Resistive Therapy Group | Sham Group | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (8.4) | 43.7 (10.7) | 42.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 18 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 18 | 18 | 36
Height [Mean (Standard Deviation); unit: centimeters] | 163.7 (6.3) | 165.3 (10.0) | 164.5 (8.2)
weight [Mean (Standard Deviation); unit: kg] | 62.0 (8.4) | 70.4 (12.8) | 66.2 (11.5)
BMI [Mean (Standard Deviation); unit: kg/m2] | 23.3 (4.0) | 25.8 (4.2) | 24.5 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Score Change
Description: The VAS is a tool used to help a person rate the intensity of certain sensations and feelings. This Outcome Measure will assess pain. This VAS is a straight horizontal line of fixed length from 0 to 10 cm with 0 cm indicating no pain and 10 cm indicating the worst pain imaginable.
Time Frame: baseline, pre-intervention and 24 hours after the last intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Capacitive-Resistive Therapy Group | Sham Group
Number analyzed (Participants) | 18 | 18
score on a scale
  pre-intervention | 5.9 (1.3) | 5.1 (1.2)
  24 hours after the last intervention | 4.1 (2.1) | 2.3 (1.8)

2. Primary Outcome: Pain Pressure Threshold (PPT) Score Change
Description: PPT is defined as the minimum force applied which induces pain. This measure has proven to be commonly useful in evaluating tenderness symptom. Higher scores mean better outcome.
Time Frame: baseline, pre-intervention and 24 hours after the last intervention
Measure: Mean (Standard Deviation); unit: N/m^2
Arm/Group | Capacitive-Resistive Therapy Group | Sham Group
Number analyzed (Participants) | 18 | 18
N/m^2
  Right Side pre-intervention | 2.0 (0.8) | 2.2 (0.5)
  Right Side 24 hours after the last intervention | 2.8 (0.9) | 3.1 (0.9)
  Left Side pre-intervention | 2.5 (1.3) | 2.4 (0.6)
  Left Side 24 hours after the last intervention | 2.8 (1.1) | 2.8 (0.8)

3. Secondary Outcome: Neck Disability Index (NDI) Score Change
Description: The Neck Disability Index (NDI) is a self-report questionnaire used to determine how neck pain affects a patient's daily life and to assess the self-rated disability of patients with neck pain. Each question has six statement, the first statement is marked the section score = 0, if the last statement is marked it = 5. Maximum score is 50 and minimum is 0. Lower scores mean better outcome.
Time Frame: baseline, pre-intervention and 24 hours after the last intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Capacitive-Resistive Therapy Group | Sham Group
Number analyzed (Participants) | 18 | 18
score on a scale
  pre-intervention | 28.0 (10.2) | 24.0 (8.4)
  24 hours after the last intervention | 19.7 (11.2) | 12.9 (10.5)

4. Secondary Outcome: Cervical Range of Motion (cROM) Change
Description: The cervical spine's range of motion is approximately 80° to 90° of flexion, 70° of extension, 20° to 45° of lateral flexion, and up to 90° of rotation to both sides.
Time Frame: baseline, pre-intervention and 24 hours after the last intervention
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | Capacitive-Resistive Therapy Group | Sham Group
Number analyzed (Participants) | 18 | 18
Degree
  Flexion ROM pre-intervention | 60 (12) | 63 (9)
  Flexion ROM 24 hours after the last intervention | 65 (9) | 66 (11)
  Extension ROM pre-intervention | 59 (11) | 70 (14)
  Extension ROM 24 hours after the last intervention | 66 (12) | 68 (14)
  Left Lateral Flexion ROM pre-intervention | 51 (12) | 49 (11)
  Left Lateral Flexion ROM 24 hours after the last i | 53 (9) | 56 (12)
  Right Lateral Flexion ROM pre-intervention | 47 (13) | 43 (9)
  Right Lateral Flexion ROM 24 hours after the last | 49 (11) | 54 (12)
  Left Lateral Rotation ROM pre-intervention | 77 (14) | 78 (10)
  Left Lateral Rotation ROM 24 hours after the last | 84 (7) | 82 (13)
  Right Lateral Rotation ROM pre-intervention | 75 (12) | 78 (12)
  Right Lateral Rotation ROM 24 hours after the last | 82 (10) | 80 (12)

5. Secondary Outcome: Short Form - 36 (SF-36) Score Change
Description: The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status and an abbreviated variant of it. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: baseline, pre-intervention and 24 hours after the last intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Capacitive-Resistive Therapy Group | Sham Group
Number analyzed (Participants) | 18 | 18
score on a scale
  Physical Functioning pre-intervention | 77 (11) | 71 (16)
  Physical Functioning 24 hours after the last inter | 80 (14) | 79 (13)
  Physical Role Functioning pre-intervention | 60 (39) | 61 (40)
  Physical Role Functioning 24 hours after the last | 71 (37) | 77 (32)
  Bodily Pain pre-intervention | 49 (12) | 54 (17)
  Bodily Pain 24 hours after the last intervention | 60 (15) | 70 (16)
  General Health Perceptions pre-intervention | 59 (20) | 59 (17)
  General Health Perceptions 24 hours after the last | 59 (20) | 68 (15)
  Vitality pre-intervention | 50 (16) | 55 (21)
  Vitality 24 hours after the last intervention | 49 (18) | 62 (15)
  Social Role Functioning pre-intervention | 70 (20) | 72 (19)
  Social Role Functioning 24 hours after the last in | 83 (19) | 81 (14)
  Emotional Role Functioning pre-intervention | 63 (20) | 63 (34)
  Emotional Role Functioning 24 hours after the last | 82 (24) | 74 (18)
  Mental Health pre-intervention | 68 (12) | 68 (20)
  Mental Health 24 hours after the last intervention | 72 (11) | 74 (13)

ADVERSE EVENTS:
Time Frame: In the study conducted between 12 December 2019 - 15 May 2020, no adverse effects were encountered before, during or after the 10 treatment sessions, an average of three weeks, process applied to patients.
Description: No side effects were seen. As in many physical therapy modalities, our study did not show any side effects. In the capacitive resistive therapy method used as a deep tissue heater, there is no side effect defined in the literature before.
Arm/Group | Capacitive-Resistive Therapy Group | Sham Group
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT04287517/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT04287517/ICF_001.pdf